CLINICAL TRIAL: NCT05081141
Title: Screening for HHV8 Infection in Solid Organ Transplantation Donors, Candidates and Recipients
Brief Title: HHV8 and Solid Organ Transplantation
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: S_OTTO
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: HHV8; HHV8 Infection; HHV8-Related Malignant Neoplasm; Kaposi Sarcoma; Lung Transplant; Complications; Liver Transplant; Complications; Kidney Transplant; Complications; Castleman Disease
Keywords: HHV8; Solid organ transplant; Lung transplant; Liver transplant; Kidney transplant; Kaposi Sarcoma; Castleman Disease
MeSH Terms: conditions — Sarcoma, Kaposi; Castleman Disease | interventions — Diagnostic Tests, Routine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- SOT Donors: Solid organ transplantation donors
  Interventions: Diagnostic Test: Diagnostic test for HHV8 exposure
- LuTx candidates and recipients: Lung transplant candidates and recipients
  Interventions: Diagnostic Test: Diagnostic test for HHV8 exposure
- LTx candidates and recipients: Liver transplant candidates and recipients
  Interventions: Diagnostic Test: Diagnostic test for HHV8 exposure
- KTx candidates and recipients: Kidney transplant candidates and recipients
  Interventions: Diagnostic Test: Diagnostic test for HHV8 exposure

INTERVENTIONS:
Diagnostic Test: Diagnostic test for HHV8 exposure — Venipuncture for blood sampling

SUMMARY:
Solid organ transplant candidates will undergo serological screening for HHV8 at time of listing and transplantation.

In the event of a recipient/donor mismatch R-/D+ or in the presence of a seropositive recipient (R+), blood levels of HHV8 DNA will be monitored together with specific IGRA for HHV8.

DETAILED DESCRIPTION:
Patients on the waiting list for solid organ transplantation will undergo serological screening for HHV8 (lytic and latent antigens) in the pre-transplant phase, both at time of listing and then at the time of transplantation; if seropositivity is found, further investigations will be performed, i.e. blood levels of HHV8 DNA and specific Elispot for HHV8.

As for donors, serological testing for HHV8 (lytic and latent antigens) will be performed.

AFTER SOLID ORGAN TRANSPLANTATION

* Patients found HHV8 seropositive in the pretransplant phase (R +), being at risk of HHV8 reactivation, will be monitored monthly in terms of viremia (HHV8 DNA) and specific IGRA for HHV8 for the first 6 months after transplantation and subsequently every 3 months up to 12 months post transplant.
* In case of patients who were found HHV8 seronegative at time of transplantation, donor serology will be evaluated. In case of R-/D+ mismatch, SOT recipients will receive the same monitoring of R + patients (blood levels of HHV8 DNA and specific IGRA for HHV8 monthly for the first 6 months and then every 3 months up to 12 months after transplantation).
* With reference to lung transplant patients, in cases of R + or R- / D +, HHV8 DNA will also be searched on the BAL obtained during surveillance bronchoscopies (usually at 3, 6 and 12 months after transplantation).

ELIGIBILITY:
SOT DONORS:

Inclusion Criteria:

* all donors used for transplantation purposes (kidney, liver, lung), including living donors in case of kidney transplantation

Exclusion Criteria:

* None

SOT CANDIDATES RECIPIENTS:

Inclusion Criteria:

* All patients listed for solid organ transplantation (lung, liver and kidney)

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will include all the donors being used for transplantation purposes at our centre and the respective recipients.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of HHV8 seropositivity among SOT donors and recipients | 2021-2024
  Incidence of HHV8 seropositivity among solid organ transplantations donors, candidates and recipients
Incidence of HHV8 mismatch between SOT donors and recipients | 2021-2024
  Incidence of HHV8 mismatch between solid organ transplantations donors and recipients

SECONDARY OUTCOMES:
Incidence of HHV8 related disease after solid organ transplantation | 2021-2025
  Incidence of HHV8 related disease after solid organ transplantation

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico di Milano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polizzotto MN, Uldrick TS, Wyvill KM, Aleman K, Marshall V, Wang V, Whitby D, Pittaluga S, Jaffe ES, Millo C, Tosato G, Little RF, Steinberg SM, Sereti I, Yarchoan R. Clinical Features and Outcomes of Patients With Symptomatic Kaposi Sarcoma Herpesvirus (KSHV)-associated Inflammation: Prospective Characterization of KSHV Inflammatory Cytokine Syndrome (KICS). Clin Infect Dis. 2016 Mar 15;62(6):730-738. doi: 10.1093/cid/civ996. Epub 2015 Dec 12. PMID 26658701
- [Background] Chiereghin A, Barozzi P, Petrisli E, Piccirilli G, Gabrielli L, Riva G, Potenza L, Cappelli G, De Ruvo N, Libri I, Maggiore U, Morelli MC, Potena L, Todeschini P, Gibertoni D, Labanti M, Sangiorgi G, La Manna G, Pinna AD, Luppi M, Lazzarotto T. Multicenter Prospective Study for Laboratory Diagnosis of HHV8 Infection in Solid Organ Donors and Transplant Recipients and Evaluation of the Clinical Impact After Transplantation. Transplantation. 2017 Aug;101(8):1935-1944. doi: 10.1097/TP.0000000000001740. PMID 28333859
- [Background] Pietrosi G, Vizzini G, Pipitone L, Di Martino G, Minervini MI, Lo Iacono G, Conaldi PG, Grossi P, Lamonaca V, Galatioto L, Gruttadauria S, Gridelli B. Primary and reactivated HHV8 infection and disease after liver transplantation: a prospective study. Am J Transplant. 2011 Dec;11(12):2715-23. doi: 10.1111/j.1600-6143.2011.03769.x. Epub 2011 Oct 3. PMID 21966899
- [Background] Riva G, Luppi M, Barozzi P, Forghieri F, Potenza L. How I treat HHV8/KSHV-related diseases in posttransplant patients. Blood. 2012 Nov 15;120(20):4150-9. doi: 10.1182/blood-2012-04-421412. Epub 2012 Sep 11. PMID 22968461
- [Background] Tzannou I, Papadopoulou A, Naik S, Leung K, Martinez CA, Ramos CA, Carrum G, Sasa G, Lulla P, Watanabe A, Kuvalekar M, Gee AP, Wu MF, Liu H, Grilley BJ, Krance RA, Gottschalk S, Brenner MK, Rooney CM, Heslop HE, Leen AM, Omer B. Off-the-Shelf Virus-Specific T Cells to Treat BK Virus, Human Herpesvirus 6, Cytomegalovirus, Epstein-Barr Virus, and Adenovirus Infections After Allogeneic Hematopoietic Stem-Cell Transplantation. J Clin Oncol. 2017 Nov 1;35(31):3547-3557. doi: 10.1200/JCO.2017.73.0655. Epub 2017 Aug 7. PMID 28783452